CLINICAL TRIAL: NCT01961089
Title: GALILEI Lens Professional vs. Predicate Devices: a Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziemer Ophthalmic Systems AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ZIOS-13/01
Record Dates: First submitted 2013-10-07; First posted 2013-10-11 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal (Experimental): Arm: Normal eyes Interventions: Galilei Lens Professional, IOLMaster, Lenstar
  Interventions: Device: Galilei Lens Professional; Device: IOLMaster; Device: Lenstar
- Mild Cataract (Active Comparator): Arm: Eyes with mild cataract Interventions: Galilei Lens Professional, IOLMaster, Lenstar
  Interventions: Device: Galilei Lens Professional; Device: IOLMaster; Device: Lenstar
- Severe cataract (Experimental): Arm: Eyes with severe cataract Interventions: Galilei Lens Professional, IOLMaster, Lenstar
  Interventions: Device: Galilei Lens Professional; Device: IOLMaster; Device: Lenstar

INTERVENTIONS:
Device: Galilei Lens Professional — Measurement device
Device: IOLMaster — Measurement device
Device: Lenstar — Measurement device

SUMMARY:
Study question: How does the new GALILEI Lens Professional compare to predicate devices? Study hypothesis: The GALILEI Lens Professional achieves a better precision in the postoperative, calculated target refraction with cataract surgeries than predicate devices, and it is more versatile in the measurable parameters as well as more user-friendly.

DETAILED DESCRIPTION:
Background: An accessory to the commercially available GALILEI Dual-Scheimpflug Corneal Topographer/Keratometer with the name "EBR Accessory" was developed by the company Ziemer Ophthalmic Systems AG for the measurement of intraocular distances. The combination is called "GALILEI Lens Professional". The measurement principle is based on on short coherence interferometry/-reflectometry, which has gained wide-spread application and has been applied clinically, including one of the members of this study group, for the precise measurement of axial, intraocular distances (12.1.). Such EBR Accessory measurements, in combination with measurements by the GALILEI, may be applied to given intra-ocular lens (IOL) types and IOL equations, an permit the calculation of suggested IOLs that are implanted during cataract surgery, in order to achieve the desired vision correction. To register this accessory for sale, the precision and agreement to existing devices with similar applications ("predicate devices") must be demonstrated. One complete measurement consists of a cornea-topography/keratometry scan, followed immediately by three consecutive, axial biometry scans of the anterior segment (cornea and crystalline lens) and - after a short re-alignment - three consecutive, axial biometry scans of the retina. The measurement process is continuous, but divided in two steps. Blinking by the patient is possible in between the two steps, which increases patient comfort and, in certain cases, measurement success. Precision is evaluated by three repeated, complete measurements with the GALILEI Lens Professional and each predicate device. Two standard devices with comparable optical technology that are used in routine cataract surgery were declared as predicate devices. These two devise are typically used in combination with standard keratometers, as which the GALILEI Lens Professional may be employed as well.

Goal: The comparison of the GALILEI Lens Professional to predicate devices with respect to precision in measuring postoperative, calculated target refractions in cataract patients, and versatility of measurable quantities.

ELIGIBILITY:
Inclusion Criteria:

* spherical equivalent between -10 D and +10 D
* best-corrected VA of 20/100 or better.

Exclusion Criteria:

* strabism
* blepharitis
* nystagmus
* amblyopia
* anisometropia (spherical equivalent > 1D)
* angle closure glaucoma
* seizure disorder
* brain damages
* Down syndrome
* trisomy 13 or 18
* cerebral palsy
* other serious disorders of the eye or central nervous systems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bojan Pajic, MD, Principal Investigator — Eye Clinic Orasis
Locations (1):
- Eye Clinic Orasis, Reinach, Canton of Aargau, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 adult subjects were recruited from among patients seen at the ORASIS eye clinics, including 20 people with cataract in at least one eye and 20 subjects without cataract. The subjects included 5 people with prior refractive surgery, 5 people with high myopia, 5 people with high hyperopia, and 3 persons with dilated pupils.
Groups:
- Device: Galilei Lens Professional versus predicate devices:
  Galilei G6 Lens Professional (Ziemer Ophthalmic Systems AG) IOLMaster (Carl Zeiss Meditech) Lenstar 900 (Haag-Streit AG)
Period: Overall Study
Arm/Group | Device
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Device: Galilei Lens Professional versus predicate devices
  Galilei G6 Lens Professional (Ziemer Ophthalmic Systems AG) IOLMaster (Carl Zeiss Meditech) Lenstar 900 (Haag-Streit AG)
Arm/Group | Device
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (18.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 11
Region of Enrollment [Number; unit: participants]
  Switzerland | 40

OUTCOME MEASURES:

1. Primary Outcome: Agreement With Predicate Devices in Terms of Agreement 1
Description: Assessed parameters:
  Axial Length (AL; G6, IOLM, LS) Central Corneal Thickness (CCT; G6, LS)) Anterior Chamber Depth (ACD; G6, IOLM, LS) Lens Thickness (LT; G6, LS) Corneal Curvature (SimK; G6, IOLM, LS) White-to-White (WtW; G6, IOL, LS)
Time Frame: 3 months
Population: The measurement of Central Corneal Thickness (CCT) and Lens Thickness (LT) is not possible with the IOLM: the IOLM cannot measure these two parameters and does therefore not display results for CCT and LT. As a consequence, the comparison in CCT and LT is only possible between the G6 and the LS, but not with respect to the IOLM.
Measure: Mean (Standard Deviation); unit: Units are mm
Units Other Than Participants: eyes
Groups:
- Device: Galilei Lens G6 Professional (G6) versus IOLMaster (IOLM) and Lenstar 900 (LS)
Arm/Group | Device
Number analyzed (Participants) | 40
Number analyzed (eyes) | 72
Units are mm
  AL G6-IOLM | -0.010 (0.049)
  AL G6-LS | -0.023 (0.048)
  AL IOLM-LS | -0.014 (0.020)
  CCT G6-LS | 0.005 (0.008)
  ACD G6-IOLM | 0.137 (0.104)
  ACD G6-LS | 0.052 (0.168)
  ACD IOLM-LS | -0.087 (0.220)
  LT G6-LS | 0.070 (0.256)
  WtW G6-IOLM | 0.150 (0.199)
  WtW G6-LS | -0.121 (0.173)
  WtW IOLM-LS | -0.276 (0.191)
Statistical Analysis 1: Comparison: Device; P-value comparing AL between G6 and IOLM; Test type: Equivalence — The significance of a difference in a measured parameter between two devices was assessed using a paired t-test; p = 0.09, Paired t-test
Statistical Analysis 2: Comparison: Device; P-value comparing AL between G6 and LS; Test type: Equivalence — The significance of a difference in a measured parameter between two devices was assessed using a paired t-test; p < 0.001, Paired t-test
Statistical Analysis 3: Comparison: Device; P-value comparing AL between IOLM and LS; Test type: Equivalence — The significance of a difference in a measured parameter between two devices was assessed using a paired t-test; p < 0.0001, Paired t-test
Statistical Analysis 4: Comparison: Device; P-value comparing CCT between G6 and LS; Test type: Equivalence — The significance of a difference in a measured parameter between two devices was assessed using a paired t-test; p < 0.0001, Paired t-test
Statistical Analysis 5: Comparison: Device; P-value comparing ACD between G6 and IOLM; Test type: Equivalence — The significance of a difference in a measured parameter between two devices was assessed using a paired t-test; p < 0.0001, Paired t-test
Statistical Analysis 6: Comparison: Device; P-value comparing ACD between G6 and LS; Test type: Equivalence — The significance of a difference in a measured parameter between two devices was assessed using a paired t-test; p < 0.01, Paired t-test
Statistical Analysis 7: Comparison: Device; P-value comparing ACD between IOLM and LS; Test type: Equivalence — The significance of a difference in a measured parameter between two devices was assessed using a paired t-test; p = 0.02, Paired t-test
Statistical Analysis 8: Comparison: Device; P-value comparing LT between G6 and LS; Test type: Equivalence — The significance of a difference in a measured parameter between two devices was assessed using a paired t-test; p < 0.01, Paired t-test
Statistical Analysis 9: Comparison: Device; P-value comparing WtW between G6 and IOLM; Test type: Equivalence — The significance of a difference in a measured parameter between two devices was assessed using a paired t-test; p < 0.0001, Paired t-test
Statistical Analysis 10: Comparison: Device; P-value comparing WtW between G6 and LS; Test type: Equivalence — The significance of a difference in a measured parameter between two devices was assessed using a paired t-test; p < 0.0001, Paired t-test
Statistical Analysis 11: Comparison: Device; P-value comparing WtW between IOLM and LS; Test type: Equivalence — The significance of a difference in a measured parameter between two devices was assessed using a paired t-test; p < 0.001, Paired t-test

2. Secondary Outcome: Agreement With Devices of the Same Type in Terms of Repeatability
Description: Assessed parameters:
  Axial Length (AL) Central Corneal Thickness (CCT) Anterior Chamber Depth (ACD) Lens Thickness (LT) Corneal Curvature (SimK) White-to-White (WtW)
Time Frame: 3 months
Population: The IOLM does not measure CCT and LT. Thus, repeatability results are available with the G6 and the LS, but not with the IOLM. The IOL Master displays one average value only for WtW, which does not permit the calculation of repeatability under the present study design.
Measure: Number; unit: Coefficient of variation
Units Other Than Participants: Eyes
Arm/Group | Device
Number analyzed (Participants) | 40
Number analyzed (Eyes) | 80
Coefficient of variation
  AL G6 | 0.0018
  AL IOLM | 0.0010
  AL LS | 0.0008
  CCT G6 | 0.0040
  CCT LS | 0.0082
  ACD G6 | 0.0259
  ACD IOLM | 0.0084
  ACD LS | 0.0391
  LT G6 | 0.0394
  LT LS | 0.0262
  SimK G6 | 0.0028
  SimK IOLM | 0.0024
  SimK LS | 0.0050
  WtW G6 | 0.0149
  WtW LS | 0.0042
Statistical Analysis 1: Comparison: Device; Repeatability was determined with random effect ANOVAs (estimates of random effects). They were calculated as the square root of the sum of the (Device x EyeID) interaction component plus (EyeID) and (Device) variance components plus the residual variance component. A (Device x Operator) interaction component was not assessed because each device was consistently operated by the same operator such that there was no Device x Operator interaction component. CV = Coefficient of Variation = SD/mean; Test type: Superiority or Other; p = 0.05, ANOVA

3. Primary Outcome: Agreement With Predicate Devices in Terms of Agreement 2
Description: Assessed Parameters:
  Simulated Corneal Curvature (SimK; G6, IOLM, LS)
Time Frame: 3 months
Population: SimK
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Device
Number analyzed (Participants) | 40
Diopters
  SimK G6-IOLM | -0.031 (0.247)
  SimK G6-LS | -0.033 (0.326)
  SimK IOLM-LS | 0.008 (0.198)
Statistical Analysis 1: Comparison: Device; P-value comparing SimK between G6 and IOLM; Test type: Equivalence — The significance of a difference in a measured parameter between two devices was assessed using a paired t-test; p = 0.13, Paired t-test
Statistical Analysis 2: Comparison: Device; P-value comparing SimK between G6 and LS; Test type: Equivalence — The significance of a difference in a measured parameter between two devices was assessed using a paired t-test; p = 0.25, Paired t-test
Statistical Analysis 3: Comparison: Device; P-value comparing SimK between IOLM and LS; Test type: Equivalence — The significance of a difference in a measured parameter between two devices was assessed using a paired t-test; p = 0.21, Paired t-test

ADVERSE EVENTS:
Time Frame: 3 months
Description: No adverse events were observed
Groups:
- Device: Galilei G6 Lens Professional versus IOLMaster and Lenstar
Arm/Group | Device
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

LIMITATIONS AND CAVEATS:
Due to the the removal and non-repetition of poor-quality G6 measurements, the informative value of the repeatability results is limited. Direct comparison to the predicates is problematic, as poor-quality measurements with those were repeated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No